CLINICAL TRIAL: NCT06396754
Title: Deployment and Clinical Evaluation of an AI-powered Digital Oncology Biomarker Tool to guidE Treatment in TNBC
Acronym: AIDOBE
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Case45 Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: CCR6030
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AI-analysis on diagnostic and surgical specimens — The analysis will report a list of AI-based biomarkers to assess the tumour-immune spatial microenvironment as well as final spatial immune-ecology prognostic (SIPA) reports for every patient.

SUMMARY:
TILs have been shown to be predictive for response to neo-adjuvant chemotherapy in patients with TNBC in multiple studies (Level-1B evidence for clinical validity as per REMARK criteria). TNBC patients with excellent survival outcome and low incidence of metastasis can be identified using a manual TIL score.

Furthermore, a fully end-to-end blinded evaluation of the same algorithm to be used in this study achieved >90% accuracy for predicting disease free survival (DFS) and overall survival (OS) in the pooled analysis of seven adjuvant phase-III TNBC trials.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Confirmed diagnosis of triple negative breast cancer (non-metastatic)
* Planned for neo-adjuvant systemic therapy
* Written consent to generic Tissue for Research donation

Exclusion Criteria:

* Patients declined consent for generic Tissue for Research donation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with triple negative breast cancer requiring neoadjuvant systemic therapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
To determine the reliability and performance of the process and AI tool | 6 months
  Success rate of digitization of H&E slides & Turnaround time for biomarker report within standard patient pathways

CONTACTS AND LOCATIONS:
Overall Officials: Navita Somaiah, Principal Investigator — Institute of Cancer Research, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided